CLINICAL TRIAL: NCT03405350
Title: Evaluation of Spa Medicine on the Example of Comprehensive Therapy in the Spa Resort Przerzeczyn Zdroj
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jadwiga Kuciel-Lewandowska, Doctor of Medicine, Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB 401/2008
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis; Degenerative Disc Disease
MeSH Terms: conditions — Osteoarthritis; Intervertebral Disc Degeneration | interventions — Laser Therapy; Cryotherapy; Electric Stimulation Therapy; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The treatment included a comprehensive therapy: redon-sulfide baths, partial mud baths, kinesiotherapy, terrain therapy, dry massage, laser therapy, low-frequency magnetic field, ultrasonotherapy, cryotherapy, electrotherapy, light therapy. On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, the concentration of endorphins and serotonin, bilirubin, uric acid, albumin) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: VAS scale and anxiety and depression levels - HADS scale.
  Interventions: Procedure: Redon-sulfide baths; Procedure: Partial Mud Baths; Procedure: Kinesiotherapy; Procedure: Terrain Therapy; Procedure: Dry Massage; Procedure: Laser Therapy; Procedure: Low-frequency Magnetic Field; Procedure: Ultrasonotherapy; Procedure: Cryotherapy; Procedure: Electrotherapy; Procedure: Light Therapy
- Control Group (No Intervention): On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, the concentration of endorphins and serotonin, bilirubin, uric acid, albumin) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: VAS scale and anxiety and depression levels - HADS scale.

INTERVENTIONS:
Procedure: Redon-sulfide baths — Encompassing whole body or isolated limbs - upper and/or lower limbs - temperature: 37-38 degrees Celsius, duration: 20 minutes.
  Arms: Study Group
Procedure: Partial Mud Baths — duration: 20 minutes, temperature 40-42 degrees Celsius
  Arms: Study Group
Procedure: Kinesiotherapy — It is the therapeutic treatment of disease by passive and active muscular movements (as by massage) and of exercise. It is the core element of physiotherapy/physical therapy. Kinesiotherapy - duration of 30-45 min.
  Arms: Study Group
Procedure: Terrain Therapy — walking, outdoors physical activities,
  Arms: Study Group
Procedure: Dry Massage — Depending on the needs of each patient it involved cervical (CC), thoracic (TH), or lumbar spine (LS).
  Arms: Study Group
Procedure: Laser Therapy — treatment parameters: sweeping, continuous, wavelength 808 nm, power 12 J, 400mV, duration 30s,
  Arms: Study Group
Procedure: Low-frequency Magnetic Field — duration 20 minutes, impulse shape - rectangular, induction 5 mT, frequency 20-50Hz,
  Arms: Study Group
Procedure: Ultrasonotherapy — treatment parameters: 800kHz/6cm2 head, ultrasound impulse wave: 2ms - impulse, 9ms - break, dose 0.5-0.6 W/cm2 over 6 minutes,
  Arms: Study Group
Procedure: Cryotherapy — ventilator, treatment duration 2-3 minutes, temperature - 80 to - 110 degrees Celsius,
  Arms: Study Group
Procedure: Electrotherapy — Bernard's diadynamic currents - treatment parameters: DF1 CP4 LP4, Nemec interference currents (frequency range 0-100Hz), percutaneous electrostimulation (TENS) - rectangular impulse currents, impulse duration 0.2ms, frequency 40Hz, regulated current 0-100mA,
  Arms: Study Group
Procedure: Light Therapy — blue filter Sollux lamp, radiation distance 30-40 cm, duration 15 minutes, Bioptron lamp - radiation distance 10 cm, duration 5-10 minutes
  Arms: Study Group

SUMMARY:
Observation conducted during the 21 days of treatment in the health resort of Przerzeczyn Zdroj. In a treatment of applied therapy: redon-sulfide baths, partial mud baths, kinesitherapy, terrain therapy, dry massage, laser therapy, low-frequency magnetic field, ultrasonotherapy, cryotherapy, electrotherapy, light therapy. Study group with joint or back pain due to osteoarthritis or degenerative disc disease. The control group was selected by the spa workers, healthy individuals, nonsmokers, who did not drink alcohol. It was recommended to retain the previous lifestyle and use of resort's facilities was prohibited. In both of these groups, appropriate pre- and post-treatment studies were performed.

DETAILED DESCRIPTION:
The observation was conducted during 21 days of medicinal stays in the health resort of Przerzeczyn Zdroj. The treatment included a comprehensive therapy: redon-sulfide baths, partial mud baths, kinesitherapy, terrain therapy, dry massage, laser therapy, low-frequency magnetic field, ultrasonotherapy, cryotherapy, electrotherapy, light therapy.

The study group consisted of patients with joint or back pain due to osteoarthritis or degenerative disc disease.participating in therapy. On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, the concentration of endorphins and serotonin, bilirubin, uric acid, albumin) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity VAS scale and anxiety and depression levels - HADS scale.

The control group was selected by the spa workers. On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, the concentration of endorphins and serotonin) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: VAS scale and anxiety and depression levels - HADS scale.

ELIGIBILITY:
Inclusion Criteria:

* the presence of degenerative disc disease and/or osteoarthritis ;
* age range 30-69 years;
* the written consent to participate in research;
* no impediment to comprehensive treatment at the spa.

Exclusion Criteria:

* the lack of consent to participate in research;
* the age under 30 and over 70 years;
* the presence of diseases constituting a contraindication to therapy (compatible with the standard list of indications and contraindications to spa therapy);

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change of results Laboratory tests (lipids profile, CRP, smear blood morphology) on day 5 and after 18 days of therapy | on day 5 and after 18 days of therapy
  The biological material was taken with sterile disposable equipment. After 10 ml of venous blood was collected in a closed system, local laboratory tests were performed, such as morphology with smear, CRP, glycemic control, and lipids profile. Tested using standard tests.
Change of results TAS- total antioxidative potential | on day 5 and after 18 days of therapy
  The biological material was taken with sterile disposable equipment. After 5 ml of venous blood was collected in the closed system directly into the monoveta was centrifuged to obtain serum - a sample to be tested for TAS. Subsequently, specimens were transported at +6 ° C. Analyzes carried out by non-standard and non-commercial laboratory tests serving exclusively for scientific research in the Department of Medical Analyzes of the Medical University of Wroclaw.
Change of results the concentration of endorphins and serotonin | on day 5 and after 18 days of therapy
  The biological material was taken with sterile disposable equipment. After 10 ml of venous blood was collected in the closed system will be left to solidify - sample for the concentration of endorphins and serotonin. Subsequently, specimens were transported at +6 ° C. Analyzes carried out by non-standard and non-commercial laboratory tests serving exclusively for scientific research in the Department of Medical Analyzes of the Medical University of Wroclaw.

SECONDARY OUTCOMES:
Pain Index | on day 5 and after 18 days
  VAS scale (The visual analogue scale) It is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. This continuous (or "analogue") aspect of the scale differentiates it from discrete scales such as the Likert scale. There is evidence showing that visual analogue scales have superior metrical characteristics than discrete scales, thus a wider range of statistical methods can be applied to the measurements.
Anxiety and Depression Index | on day 5 and after 18 days
  HADS scale (Hospital Anxiety and Depression Scale) It was originally developed by Zigmond and Snaith (1983)and is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Zigmond and Snaith created this outcome measure specifically to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness, for example fatigue and insomnia or hypersomnia. This, it was hoped, would create a tool for the detection of anxiety and depression in people with physical health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Kuciel-Lewandowska, MD, Study Director — MD, Departament of Spa Treatment, History Physical Medicine and Balneology Medical University of Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided
Any request to share the IPD will be considered individually and in the group of all researchers who have participated in the research.

REFERENCES:
- [Derived] Kuciel-Lewandowska J, Kasperczak M, Paprocka-Borowicz M. Assessment of Changes in the Hemoglobin Level under the Influence of Comprehensive Spa Therapy Using Therapeutic Radon-Sulfur Waters and Its Correlation with Free Radical Reactions. Evid Based Complement Alternat Med. 2020 Jul 20;2020:4637129. doi: 10.1155/2020/4637129. eCollection 2020. PMID 32774419
- [Derived] Kuciel-Lewandowska J, Kasperczak M, Lewandowski LB, Paprocka-Borowicz M. Assessment of the Level of Pain Intensity and the Level of Anxiety Treated as State and Trait in Patients with Osteoarthritis of the Limbs. Pain Res Manag. 2020 Apr 23;2020:5904743. doi: 10.1155/2020/5904743. eCollection 2020. PMID 32377287
- [Derived] Kuciel-Lewandowska J, Kasperczak M, Bogut B, Heider R, Laber WT, Laber W, Paprocka-Borowicz M. The Impact of Health Resort Treatment on the Nonenzymatic Endogenous Antioxidant System. Oxid Med Cell Longev. 2020 Jan 31;2020:8423105. doi: 10.1155/2020/8423105. eCollection 2020. PMID 32089783